CLINICAL TRIAL: NCT00726973
Title: A Pilot Study With Reduced Fluence Photodynamic Therapy With Visudyne Ranibizumab VS. Ranibizumab Only to Treat Exudative AMD
Brief Title: Pilot Study Reduced Fluence PDT /Visudyne With Ranibizumab vs Ranibizumab Monotherapy for Exudative Age-related Macular Degeneration (AMD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit study participants
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-085
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Macular Edema
Keywords: Macular edema
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Reduced fluence (3300mW/cm2-50% standard fluence) PDT + ranibizumab
  Interventions: Drug: Ranibizumab
- 2 (Active Comparator): Ranibizumab monotherapy
  Interventions: Drug: Ranibizumab monotherapy

INTERVENTIONS:
Drug: Ranibizumab — Ranibizumab, and reduced fluence PDT or sham PDT and Ranibizumab. For 2 months injected intravitreal Ranibizumab will be given. At month 3 subjects will receive combination reduced fluence PDT and intravitreal Ranibizumab. If they develop recurrence of subretinal fluid, cystoid macular edema, increased pigment epithelial detachment (PED), or increased retinal thickness >100 microns compared to best thickness measure of OCT, subjects will be eligible for repeat combination reduced fluence PDT + intravitreal Ranibizumab every 3 months thereafter.
  Other Names: Lucentis
  Arms: 1
Drug: Ranibizumab monotherapy — 3 monthly intravitreal injections of Ranibizumab monotherapy. After month 2 they are eligible for retreatment with Ranibizumab if retreatment criteria are met (same as arm 1) At intervals of no less than 3 months from the previous sham PDT they will receive sham PDT if retreatment criteria are met.
  Other Names: lucentis
  Arms: 2

SUMMARY:
The purposes of this study is to determine if combination reduced fluence photodynamic therapy and Ranibizumab has:

Similar efficacy to Ranibizumab (Lucentis) alone. The ability to reduce the number of intravitreal injection of Ranibizumab or a 13 month period The ability to reduce the number of PDT treatments. The study will also collect information on the safety of combination therapy and single therapy.

DETAILED DESCRIPTION:
This will be a 13 month prospective, blinded, randomized sham controled parallel safety study. There will be 2 treatment arms.

Arm 1 will receive reduced fluence PDT at baseline followed immediately by an intravitreal injection of Lucentis. Subjects in arm 1 will receive 2 additional injections of Ranibizumab (Lucentis) over the next 2 months. Starting at month 3, they will receive combination reduced fluence PDT and intravitreal Ranibizumab (Lucentis) if they develop recurrence of the subretinal fluid, cystoid macular edema, increased pigment epithelial detachment (PED), or increased retinal thickness > 100 microns compared to the best prior thickness measure on OCT. Patients will be eligible for repeat combination reduced fluence PDT + intravitreal Ranibizumab (Lucentis) every 3 months thereafter. Group 1 patients are eligible for treatment with combination reduced fluence PDT and Ranibizumab (Lucentis) at any point at the 3 month time point or thereafter. After month 3, if patients were not eligible for combined therapy (<3 months since the last combination therapy) and have >2 lines of vision loss or > 100 microns of increased retinal thickness on OCT compared to most recent measure at their monthly visit, they would be eligible for an injection of Ranibizumab (Lucentis) as monotherapy. Thereafter, subjects will have combination therapy if retreatment criteria were met and it has been >3 months since the last PDT treatment.

Study arm 2 will receive 3 monthly intravitreal injections of Ranibizumab (Lucentis). Following month 2, they will be eligible for re-treatment with Ranibizumab (Lucentis) if retreatment criteria are met (same criteria as study arm 1). At intervals of no less than 3 months from the previous sham PDT, they will receive sham PDT if retreatment criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Male / Female > 50 years of age
* FA diagnosis of CNV lesions as described above
* Have a best corrected visual acuity letter score in the study eye between 72-24 letters (approximately 20/40 to 20/320) using ETDRS chart measured at 4 meters
* Central retinal (including lesion) thickness greater than or equal to 250 microns as measured by OCT
* Subretinal hemorrhage making up less than 50% of total lesion size and sparing the fovea
* Sufficiently clear ocular media including the lens to allow photography of the retina
* Written informed consent has been obtained.

Exclusion Criteria:

* Dense subfoveal hemorrhage (>50% of the lesion)
* Tear or rip of the retina pigment epithelium, idiopathic parafoveal telangiectasis or serous pigment epithelial detachment without CNV
* Geographic atrophy involving the foveal center
* Subretinal fibrotic scar in the study eye greater than 25% of the lesion
* Presence of any condition in study eye other than AMD known to be associated with CNV
* History diabetic retinopathy or diabetic macular edema
* Previous pars plana vitrectomy
* Previous photodynamic therapy in the study eye
* Previous photodynamic therapy in the fellow eye with resultant choroidal hypoperfusion
* Previous intravitreal anti-VEGF or steroid injection in the study eye
* Previous thermal subfoveal laser treatment in study eye
* Anticipated need for ocular surgery in the study eye during the 13 month study period
* Known allergy or sensitivity to the study medication(s) its components, diagnostic agents used during the study (Fluorescein, dilation drops) or other agents required for the study procedures (ie: povidone iodine)
* Porphyria or other porphyrin sensitivity

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy will be proportion of subjects with best corrected visual acuity improvement of 15 or more letters from baseline and wil visual acuity stabilization, less than 15 letter loss from baseline at 13 months | at conclusion of subject enrollment

SECONDARY OUTCOMES:
Mean change in ETDRS from baseline, number of Ranibizumab treatments w/reduced fluence PDT, proportion of patients with 6 lines of vision loss | at conclusion of subject enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Marx, M.D., Principal Investigator — Lahey Clinic Medical Center